CLINICAL TRIAL: NCT06843395
Title: Assessing the Feasibility, Acceptability and Effectiveness of an Transdiagnostic Acceptance and Commitment Therapy-based Ecological Momentary Intervention in College Students: a Pilot Randomized Controlled Trial
Brief Title: ACT-based EMI in College Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSEARS20250214003
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants Study

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mood monitoring condition (Placebo Comparator): Only pre- and post-assessments and ecological momentary assessment (EMA) measurements are conducted.
  Interventions: Other: Mood monitoring
- ACT-based EMI group (Experimental): Participants are required to complete a 7-day ecological momentary intervention (EMI).
  Interventions: Behavioral: ACT-based ecological momentary intervention

INTERVENTIONS:
Behavioral: ACT-based ecological momentary intervention — The intervention is based on Acceptance and Commitment Therapy (ACT) and includes the six core processes (being present, acceptance, defusion, self-as-content, values, and taking action). It is delivered in the form of an ecological momentary intervention (EMI), lasting for 7 days with two sessions per day. The intervention aims to enhance mental health, well-being, and psychological flexibility.
  Arms: ACT-based EMI group
Other: Mood monitoring — Participants do not receive any intervention. During the intervention period, they only need to complete ecological momentary assessments twice a day.
  Arms: Mood monitoring condition

SUMMARY:
This study aims to evaluate the acceptability and effectiveness of a transdiagnostic, Acceptance and Commitment Therapy (ACT)-based ecological momentary intervention (EMI) among college students. A mixed-methods pilot randomized controlled trial (RCT) will be conducted to assess its impact on psychological flexibility, well-being and mental health outcomes.

DETAILED DESCRIPTION:
Mental health issues are prevalent among college students, yet traditional interventions often face barriers related to accessibility and engagement. This study explores the feasibility, acceptability, and preliminary effectiveness of a transdiagnostic ACT-based EMI designed to deliver in-the-moment psychological support via digital platforms. A mixed-methods pilot RCT will be conducted, with participants randomly assigned to either the ACT-based EMI group or a mood monitoring group. Quantitative measures will assess changes in psychological flexibility, stress, anxiety, depression, and well-being, while qualitative interviews will provide insights into user experience, engagement, and perceived benefits or barriers. Findings from this study will inform the optimization of ACT-based digital interventions for college students and contribute to the growing field of personalized, technology-assisted mental health care.

ELIGIBILITY:
Inclusion Criteria:

* Participants in our study are healthy college students
* have smartphone, and have access to the internet

Exclusion Criteria:

* currently participating in another research
* have significant cognitive impairment that prevents participation in the research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall mental health | Baseline (pre-intervention); Immediately after the intervention (1 week after baseline); 1-month follow-up (1 month after intervention)
  Overall mental health will be measured using the 12-item General Health Questionnaire (GHQ-12). Each item is rated on a 4-point Likert scale, with total scores ranging from 0 to 36. Higher scores indicate greater mental health difficulty.
Psychological distress | Baseline (pre-intervention); Immediately after the intervention (1 week after baseline); 1-month follow-up (1 month after intervention)
  Psychological distress will be measured using the 21-item Depression Anxiety Stress Scale. They ask about depressive symptoms, anxiety symptoms, and general stress symptoms. Each item is rated on a 4-point Likert scale from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). Higher scores indicate more psychological distress
Mental well-being | Baseline (pre-intervention); Immediately after the intervention (1 week after baseline); 1-month follow-up (1 month after intervention)
  The 14-item Mental Health Continuum-Short Form (MHC-SF) will be used to measure mental well-being during the past month. This scale has 3 dimensions: emotional well-being (EWB), psychological well-being (PWB), and social well-being (SWB). Each item is rated on a 6-point scale from 0 (never) to 5 (every day), with a higher score indicating greater well-being.
Psychological flexibility and inflexibility | Baseline (pre-intervention); Immediately after the intervention (1 week after baseline); 1-month follow-up (1 month after intervention)
  The multidimensional psychological flexibility inventory short form (MPFI-24) is a 24-item scale assessing psychological flexibility. The scale consists of a flexibility subscale and an inflexibility subscale, divided into 12 dimensions, with 2 entries for each dimension, a total of 24 entries, and scored at levels 1 (never true) to 6 (always true).
Acceptability | post-intervention (one week after baseline)
  The 8-item Client Satisfaction Questionnaire (CSQ-8) is employed to measure client satisfaction. Each item is rated on a 4-point Likert scale. Higher scores reflect better client satisfaction.

SECONDARY OUTCOMES:
State anxiety and depression | During the 7-day intervention period, measurements are conducted twice per day.
  State anxiety and depression will be measured with the four-item Patient Health Questionnaire for Depression and Anxiety (PHQ-4). Responses are scored as 0 ("not at all"), 1 ("several days"), 2 ("more than half the days"), or 3 ("nearly every day"), with the total score on this composite measure ranging from 0 to 12.
State stress | During the 7-day intervention period, measurements are conducted twice per day.
  State stress will be measured using a single item adapted from the Psychological Stress Measure (PSM-9). Participants will rate their state stress level on a sliding scale from 0 (not stressed at all) to 100 (very stressed), with higher scores indicating greater perceived stress.
State well-being | During the 7-day intervention period, measurements are conducted twice per day.
  State well-being will be measured with one item inspired by the Well-Being Manifestations Measure Scale using a sliding scale ranging from 0 (not good at all) to 100 (very good).
State subjective happiness | During the 7-day intervention period, measurements are conducted twice per day.
  State subjective happiness will be measured by the 2-item Subjective Happiness Scale with each item rated on a 7-point Likert scale from 1 (not a very happy person) to 7 (a very happy person).
State affect | During the 7-day intervention period, measurements are conducted twice per day.
  State affect will be tapped by the 9-item Emmons Mood Indicator. Participants indicate their momentary feelings on a 7-point Likert scale ranging from 1 (not at all) to 7 (extremely), for NA (e.g., depressed, worried/anxious, and unhappy) and PA (e.g., joyful, happy, and enjoyment/fun).
State psychological flexibility | During the 7-day intervention period, measurements are conducted twice per day.
  State psychological flexibility will be measured with Psy-Flex, a short self-report measure which covers all aspects of psychological flexibility. Items are rated on a scale from 5 ("very often") to 1 ("very rarely") and then summed. The score is then inter-preted such that higher scores represent higher psychological flexibility.
State psychological inflexibility | During the 7-day intervention period, measurements are conducted twice per day.
  State psychological inflexibility will be measured with six item adapted from the Multidimensional psychological flexibility inventory using a sliding scale ranging from 1 (never true) to 6 (always true).
State suicide ideation | During the 7-day intervention period, measurements are conducted twice per day.
  State suicide ideation will be assessed using a single item. Participants will respond on a 0 to 4 scale, with higher scores indicating greater suicidal ideation.
Suicide ideation | Baseline (pre-intervention); Immediately after the intervention (1 week after baseline); 1-month follow-up (1 month after intervention)
  Suicide ideation will be measured using the 5-item Beck Scale for Suicide Ideation (BSS-5). Each item is rated on a three-point scale, with higher scores indicating greater suicidal ideation.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China